CLINICAL TRIAL: NCT06250270
Title: Effects of Casein Protein on Metabolism When Taken Prior to Sleep and in the Morning
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ohio University (Other)
Responsible Party: Principal Investigator, Angela Hillman, Assistant Professor, Ohio University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 22-F-7
Record Dates: First submitted 2024-01-31; First posted 2024-02-09 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Metabolism
Keywords: Metabolism
MeSH Terms: interventions — Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Blinded pre-made packets of protein or placebo with sample coding in a sealed envelope until the end of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- PRO pm, PRO am (Experimental): Participants arrive to the lab, complete 30 mins resting metabolic rate assessment. Then they are provided with a shake to drink 30 mins before bed. They return to the lab the following morning for 30 min RMR, drink another shake and do 30 mins RMR before leaving the lab.
  Interventions: Dietary Supplement: protein or placebo
- PRO pm, PLAC am (Experimental): Participants arrive to the lab, complete 30 mins resting metabolic rate assessment. Then they are provided with a shake to drink 30 mins before bed. They return to the lab the following morning for 30 min RMR, drink another shake and do 30 mins RMR before leaving the lab.
  Interventions: Dietary Supplement: protein or placebo
- PLAC pm, PRO am (Experimental): Participants arrive to the lab, complete 30 mins resting metabolic rate assessment. Then they are provided with a shake to drink 30 mins before bed. They return to the lab the following morning for 30 min RMR, drink another shake and do 30 mins RMR before leaving the lab.
  Interventions: Dietary Supplement: protein or placebo
- PLAC pm, PLAC pm (Placebo Comparator): Participants arrive to the lab, complete 30 mins resting metabolic rate assessment. Then they are provided with a shake to drink 30 mins before bed. They return to the lab the following morning for 30 min RMR, drink another shake and do 30 mins RMR before leaving the lab.
  Interventions: Dietary Supplement: protein or placebo

INTERVENTIONS:
Dietary Supplement: protein or placebo — casein protein (30g) or placebo (maltodextrin, 30g)

SUMMARY:
The purpose of this study is to investigate the effect of casein protein consumption both prior to sleep as well first thing in the morning on metabolism (increase satiety and appetite, lower resting metabolic rate, and lower blood sugar levels), when compared to nighttime protein or placebo consumption alone. Protein itself is a macronutrient that not only helps the body repair itself, and play a critical role in growth, it also aids in increasing satiety and decreasing appetite. Casein protein specifically is slow digesting dairy protein which may impact the body's metabolism for a longer period than other dairy proteins such as whey. The literature demonstrates nighttime protein ingestion prior to sleep increases metabolic rate and satiety the next morning. However, there appears to be no data on the metabolic effects of protein ingested both at night and in the morning.

ELIGIBILITY:
Inclusion Criteria:

* male
* aged 18-30

Exclusion Criteria:

* lactose intolerant
* having known sleep issues
* being on a schedule that is not uniform week to week
* those who do not eat animal-based diets
* any known or suspected food allergies
* any known health conditions (cardiovascular disease, IBS, high blood pressure, diabetes, crohn's disease)
* those that have disordered eating
* unwillingness to take blood sugar four times a day
* being a female

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — male
Enrollment: 15 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
resting metabolic rate | baseline, during the intervention
  indirect calorimetry to measure oxygen consumption (V02) and respiratory quotient (RQ)
blood glucose | baseline, during the intervention
  fasting and pre-meal blood glucose

SECONDARY OUTCOMES:
dietary intake | during the intervention
  food logs used to track food intake during all trial visits

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio University Exercise Physiology Lab, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: No